CLINICAL TRIAL: NCT05161416
Title: Comparison of the Effects of Cartoon Watching and Bubble Blowing as Distraction Methods During Venipuncture on Pain, Fear, and Anxiety in Children Aged 6-8 Years: A Randomized Experimental Study
Brief Title: The Effects of Cartoon Watching and Bubble Blowing as Distraction Methods During Venipuncture on Pain, Anxiety, and Fear in Children Aged 6-8 Years
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Guzide UGUCU, Principal Investigator, Mersin University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MersinU*GUGUCU_001
Record Dates: First submitted 2021-12-05; First posted 2021-12-17 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Pain; Anxiety; Fear; Child, Only
Keywords: Nursing; Pain Management; Distraction; Children
MeSH Terms: conditions — Pain; Anxiety Disorders; Agnosia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The children and their parents were blinded to the groups. The principal researchers (R2, R3) were blinded to the research hypotheses. Data entry researchers (R4, R5, R6) were blinded (masked) to both research hypotheses and intervention groups. Data entries (R4, R5) were performed using the codes A and B, and shared with the researchers (R1, R7, R8) after statistical analyses were conducted and the research report was written.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bubble Group (Experimental): The children started to blow bubbles 3 minutes before the procedure. The procedure and the bubble blowing intervention were terminated simultaneously.
  Interventions: Behavioral: Bubble Blowing
- Cartoon Group (Experimental): The children started to watch the cartoon 3 minutes before the procedure. The children were supported by their parents in holding the tablet. The procedure and the cartoon watching intervention were terminated simultaneously.
  Interventions: Behavioral: Cartoon Watching

INTERVENTIONS:
Behavioral: Bubble Blowing — Active Distraction Methods
  Arms: Bubble Group
Behavioral: Cartoon Watching — Passive Distraction Methods
  Arms: Cartoon Group

SUMMARY:
Active and passive distraction methods are frequently used in the nursing management of procedural pain in children. There are no studies comparing the effects of cartoon watching (passive) and bubble blowing (active) as distraction methods on pain, anxiety, and fear associated with venipuncture in children.

This study aimed to compare the effects of bubble blowing (active distraction) and cartoon watching (passive distraction) techniques on pain, anxiety, and fear during venipuncture in children aged 6-8 years.

DETAILED DESCRIPTION:
Research Hypotheses H1a= There is a difference in the mean WB-FACES score during the procedure between the bubble group (BG) and the cartoon group (CG).

H1b= There is a difference in the mean WB-FACES score after the procedure between the BG and CG groups.

H2a= There is a difference in the mean CSA score during the procedure between the BG and CG groups.

H2b= There is a difference in the mean CSA score after the procedure between the BG and CG groups.

H3a= There is a difference in the mean CFS score during the procedure between the BG and CG groups.

H3b= There is a difference in the mean CFS score after the procedure between the BG and CG groups.

Design and Settings: This parallel-group randomized trial was conducted at the invasive procedure room of the pediatrics department of a university hospital in the East Mediterranean Region of Turkey. For this experimental research, 56 children aged 6-8 years were assigned to two groups (Bubble Group=BG; n = 28 and Cartoon Group=CG; n = 28) using block randomization.

Sample Size: The main trial sample was calculated based on the pilot study findings. The pilot study was conducted with 20 children (BG; n = 10 and CG; n = 10) who met the eligibility criteria. A priori power analysis was performed based on the effect size (d = 0.885, large effect) of the difference in pain scores between the groups (during the procedure) determined in the pilot study. Using G*Power 3.1.9.7, the minimum sample size was calculated as 56 children, with 28 children per group, for a two-tailed hypothesis, an effect size of d = 0.885, an allocation ratio of n1/n2=1, type I error of 0.05, and a power of 90%.

Randomization: Using block randomization, six different combinations of the codes A and B with a block size of 4 (ABAB(1), AABB(2), BABA(3) …) were generated. The combinations were numbered from 1 to 6. The numbers (1-6) were randomly sorted 14 times via randomizer.org and a random allocation sequence was generated. Coin flipping was used to determine which of the codes A and B would be BG and CG (R1). The random allocation sequence, which was placed in opaque envelopes by giving a sequence number, was hidden from the principal researchers (R2, R3) (allocation concealment). The opaque envelopes were stored in a locked cabinet by the researcher who performed the randomization (R1). The group including the eligible children was not shared with R2 and R3 until the intervention.

Data Collection Tools Socio-Demographic Data Collection and Procedure Follow-up Form: It includes "age, gender, previous experience of hospitalization, experience of procedural pain in last week, analgesic administration at least six hours before the procedure, size of peripheral IV needle, area of IV blood sample, parental presence during procedure, and baseline data of pain, anxiety and fear scores of children before procedure".

The Wong-Bakers FACES® Pain Rating Scale (WB-FACES): Developed by Wong and Baker in 1981 and revised in 1983, the instrument is used to assess physical pain in people who are communicative, responsive, and aged three years and older. The scale consists of faces ranging from "Face 0= no hurt" to "Face 10=hurts worst".

The Children's State Anxiety Scale (CSA): Developed by Ersig et al. (2013), the Turkish validity-reliability study of this visual scale was conducted by Özalp-Gerçeker et al. (2018) and it is scored from 0 to 10. Higher values represent higher anxiety.

The Children's Fear Scale (CFS): The instrument assessed the pain-associated fear in children. Developed by McMurty et al. (2011), the Turkish validity-reliability study of this visual scale was conducted by Özalp-Gerçeker et al. (2018) and it is scored from 0 to 4. It ranges from a no fear (neutral) face (0) on the far left to a face showing extreme fear on the far right. Higher scores mean a worse outcome.

Bubble Blowing Toy: In the bubble blowing group, a two-piece toy was used that had a chamber containing diluted liquid soap, a pattern of cartoon characters and a special apparatus to generate bubbles when blown.

iPad mini: In the cartoon watching group, an iPad mini was used that had a (7.9 inch (diagonal) LED-backlit Multi-Touch display, 2048 x 1536 resolution with a density of 326 pixels per inch (ppi) with internet access.

Interventions: The invasive procedure room in the clinic was decorated with cartoon characters and ornaments on the walls. The intervention can be administered to only one child at a time in the room. In routine practice, the parental presence is supported during all invasive procedures performed on children. However, the nurses' uniforms have a print/pattern of cartoon characters in the routine practice. The room had the same characteristics for all children and their parents in terms of environmental conditions such as light, temperature, noise, and seat. Before the procedure, children's pain, anxiety, and fear were assessed after providing developmentally appropriate information. The parents were also informed about how to support their children. The same researchers performed the venipuncture (R2) and observational pain, anxiety, and fear assessments (R3) in all children. R2 and R3 are nurses with more than five years of experience in pediatrics and degrees in scientific fields.

Bubble Blowing: First, the physical comfort of the children was ensured in the invasive procedure room. Then, the children were instructed to take a deep breath through the nose and generate bubbles by slowly blowing into the special apparatus. The children's questions about the procedure and the process were answered in a developmentally appropriate manner. The children were allowed to choose a bubble blowing toy according to the printed cartoon characters. The children were supported by their parents in holding the chamber of the toy. The children started to blow bubbles 3 minutes before the procedure. The procedure and the bubble blowing intervention were terminated simultaneously. The bubble blowing toy was given to the children as a gift after the intervention.

Cartoon Watching: In the cartoon watching group, the cartoons that the children liked to watch were learned from the parents before the procedure. First, the physical comfort of the children was ensured in the invasive procedure room. The children were asked which cartoon they wanted to watch before the procedure. They started to watch the cartoon 3 minutes before the procedure. The children were supported by their parents in holding the tablet. The procedure and the cartoon watching intervention were terminated simultaneously.

Statistical Methods: The study data were analyzed using the statistical package for Social Sciences. The level of statistical significance was set at 0.05. The normality of the data was determined by the kurtosis and skewness coefficients, revealing that the scale scores were normally distributed. The data were presented as mean, standard deviation, confidence interval, frequency, and percentages. The similarities of demographic and clinical characteristics between the groups were analyzed by the Chi-square test. The mean scale scores of the groups were compared using the Independent Samples t-test.

Ethical Considerations: The study was granted approval by the clinical research ethics committee and written institutional permission by the hospital. Parents were informed about the procedure and that they could withdraw from the study at any time without explanation. Parents provided written consent and children verbal consent before the study.

ELIGIBILITY:
Inclusion Criteria:

* Child aged 6-8 years
* Child with need or plan for venipuncture (antecubital fossa)

Exclusion Criteria:

* Child with a neurodegenerative disease, mental retardation, vision and hearing problems, chronic, life-threatening (sepsis, shock, respiratory / cardiac arrest) or genetic disease
* Child with use of opioids, narcotics, analgesics or sedatives in the last 24 hours before the procedure

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 56 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2020-03-02 (Actual); Study Completion 2020-03-02 (Actual)

PRIMARY OUTCOMES:
Pain assesed by Wong-Baker FACES | Procedure (during the venipuncture)
  The Wong-Baker FACES (WB-FACES) Pain Rating Scale used. This scale uses in children aged 3 and older to rate pain severity. This numeric rating scale ranges from 0 to 10. Faces show emotions from smiling (0 = very happy/ no pain) to crying (10 = hurts worst).
Anxiety assesed by Children's State Anxiety Scale | Procedure (during the venipuncture)
  The Children's State Anxiety Scale assesses children's anxiety. This scale is drawn like a thermometer with a bulb at the bottom and also includes horizontal lines at intervals going up to the top (0-10). This scale ranges from 0 to 10. Higher values represent higher anxiety.
Fear by Children's Fear Scale | Procedure (during the venipuncture)
  The Child Fear Scale was used.This one-item scale measures procedure-related fear in children, consists of five sex-neutral faces, ranges from 0 (no fear) to 4 (extreme fear). Higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Pain assesed by Wong-Baker FACES | After procedure (at 3rd minutes after the venipuncture)
  The Wong-Baker FACES (WB-FACES) Pain Rating Scale used. This scale uses in children aged 3 and older to rate pain severity. This numeric rating scale ranges from 0 to 10. Faces show emotions from smiling (0 = very happy/ no pain) to crying (10 = hurts worst).
Anxiety assesed by Children's State Anxiety Scale | After procedure (at 3rd minutes after the venipuncture)
  The Children's State Anxiety Scale assesses children's anxiety. This scale is drawn like a thermometer with a bulb at the bottom and also includes horizontal lines at intervals going up to the top (0-10). This scale ranges from 0 to 10. Higher values represent higher anxiety.
Fear by Children's Fear Scale | After procedure (at 3rd minutes after the venipuncture)
  The Child Fear Scale was used.This one-item scale measures procedure-related fear in children, consists of five sex-neutral faces, ranges from 0 (no fear) to 4 (extreme fear). Higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Mersin University Hospital, Mersin, Yenişehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available due to ethical considerations.

REFERENCES:
- [Result] Ugucu G, Akdeniz Uysal D, Guzel Polat O, Artuvan Z, Polat Kulcu D, Aksu D, Gulgun Altintas M, Cetin H, Orekici Temel G. Effects of cartoon watching and bubble-blowing during venipuncture on pain, fear, and anxiety in children aged 6-8 years: A randomized experimental study. J Pediatr Nurs. 2022 Jul-Aug;65:e107-e114. doi: 10.1016/j.pedn.2022.03.016. Epub 2022 Apr 8. PMID 35410736